CLINICAL TRIAL: NCT02079090
Title: Ketofol Versus Fentofol for Procedural Sedation of Children 3 to 17 Years Old: a Double-Blind Randomized Controlled Trial
Brief Title: Ketofol Versus Fentofol for Procedural Sedation in the Pediatric Emergency Department
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Child and Family Research Institute (Other)
Responsible Party: Principal Investigator, Vikram Sabhaney, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H14-00273
Record Dates: First submitted 2014-03-01; First posted 2014-03-05 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Emergency Department Procedural Sedation; Fracture Reduction
Keywords: Propofol; Ketamine; Fentanyl; Procedural sedation; children; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketofol (Active Comparator): Patient will receive 0.5 mg/kg Ketamine, and 2 minutes later receive 1 mg/kg Propofol.
  Interventions: Drug: Ketofol
- Fentofol (Experimental): Patient will receive 1 microgram/kg Fentanyl, and 2 minutes later receive 1 mg/kg Propofol.
  Interventions: Drug: Fentofol

INTERVENTIONS:
Drug: Ketofol — 0.5 mg/kg Ketamine IV, and 2 minutes later receive 1 mg/kg Propofol (Diprivan).
  Arms: Ketofol
Drug: Fentofol — 1 microgram/kg Fentanyl, and 2 minutes later receive 1 mg/kg Propofol (Diprivan)
  Arms: Fentofol

SUMMARY:
Sedation and pain medication is required when bone fractures need to be fixed in the emergency department (ED). Many drugs have been used safely as single agents or in combination for the sedation of children. These drugs include Propofol, Ketamine and Fentanyl. However each of these medications has side effects and drawbacks. The combination of Propofol and Fentanyl (Fentofol) has never been compared directly with the combination of Propofol and Ketamine (Ketofol) for painful procedures in the ED, and the goal of this study is to determine which combination works better. The primary outcome of this study is to determine which drug combination has a shorter time from onset of sedation to full recovery. The investigators hypothesize that Fentofol will have shorter sedation to recovery times.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to compare the duration of procedural sedation and analgesia (PSA) from time of medication delivery to recovery for children in the ED provided by Fentofol and Ketofol.

Hypothesis: The hypothesis is that Fentofol will have a shorter duration of sedation time as compared to Ketofol.

Justification: PSA for children is a common occurrence in the ED and has been performed using Ketamine or Propofol. Propofol offers several advantages over Ketamine, including shorter recovery times, and low rates of nausea and vomiting. Propofol is a potent sedative-hypnotic that does not provide analgesia, hence another agent is commonly used in combination for painful procedures. Propofol has been used in combination with Ketamine (Ketofol) and with Fentanyl (Fentofol) to improve the quality of sedation for painful procedures such as fracture reduction. Ketofol has been shown in a double blind randomized controlled trial to be at least equivalent, or even superior to Ketamine in children who are undergoing PSA, with shorter duration of sedation, increased provider and patient satisfaction, and reduced frequency of nausea/vomiting events. A combination of 1 to 2 microgram/kg Fentanyl and 1 mg/kg Propofol has been shown to substantially reduce recovery time as compared to 0.05 mg/kg Midazolam and 1 to 2 mg/kg Ketamine, and provided adequate levels of analgesia during PSA. As a result, both Ketofol and Fentofol are considered standard treatments for PSA in the ED. However, there is currently no pediatric literature available comparing Ketofol and Fentofol for PSA in the ED setting and the results of this study will potentially identify which of the two sedation agents is superior.

ELIGIBILITY:
Inclusion Criteria:

* Children 3-17 years of age
* Presenting to the ED for assessment of a long bone fracture
* Require PSA for closed reduction of the fracture
* American Society of Anesthesia Grade I or II

Exclusion Criteria:

* Families not providing informed consent (or assent where appropriate)
* Families unable to communicate in English
* Children sustained life- or limb-threatening injuries
* Children involved in a multi-system trauma
* Children with a pathological fractures
* Children with a contraindication to using Propofol, Ketamine or Fentanyl:

Allergy or previous adverse reaction to study drugs Psychosis/schizophrenia Active upper respiratory tract infection or asthma, or chronic respiratory illnesses Coronary artery disease, congestive heart failure, hypertension, or chronic cardiac disease Chronic renal disease Increased intracranial pressure Porphyria or thyroid disorder

* Severe developmental delay or autism

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Duration of Sedation | Less than 30 minutes
  Duration of sedation is measured from time of administration of Propofol (time 0) to recovery being achieved.

SECONDARY OUTCOMES:
Recovery Time | Less than 30 minutes
  Measured from time of last dose of study drug administered to recovery
Additional analgesia or sedation medications | Less than 30 minutes
  Use of additional analgesic agents and sedation medications to complete PSA
Efficacy of sedation for completion of procedure | Less than 30 minutes
  A sedation is considered efficacious if: the patient does not have unpleasant recall of the procedure, the patient did not experience sedation-related adverse events resulting in abandonment of the procedure/permanent complication/unplanned admission to the hospital or ED, and the patient did not actively resist the procedure or require restraints.
Satisfaction with sedation | Less than 60 minutes
  Satisfaction scores will be completed by the physician performing the sedation, the physician performing the procedure, the nurse performing the sedation and by the patient in the ED. This outcome will by measured using a 5-point Likert scale, except in children between ages 6 and 9, where a 5-point facial hedonic scale is used.
Incidence of adverse events | From initiation of PSA until 48 to 72 hours post-ED discharge
  Adverse events, interventions and outcomes will be measured using the "Quebec Guidelines".

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Sabhaney, MD, Principal Investigator — University of British Columbia, BC Children's Hospital
Locations (1):
- University of British Columbia: BC Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Green SM, Roback MG, Kennedy RM, Krauss B. Clinical practice guideline for emergency department ketamine dissociative sedation: 2011 update. Ann Emerg Med. 2011 May;57(5):449-61. doi: 10.1016/j.annemergmed.2010.11.030. Epub 2011 Jan 21. PMID 21256625
- [Background] Mallory MD, Baxter AL, Yanosky DJ, Cravero JP; Pediatric Sedation Research Consortium. Emergency physician-administered propofol sedation: a report on 25,433 sedations from the pediatric sedation research consortium. Ann Emerg Med. 2011 May;57(5):462-8.e1. doi: 10.1016/j.annemergmed.2011.03.008. PMID 21513827
- [Background] Andolfatto G, Willman E. A prospective case series of pediatric procedural sedation and analgesia in the emergency department using single-syringe ketamine-propofol combination (ketofol). Acad Emerg Med. 2010 Feb;17(2):194-201. doi: 10.1111/j.1553-2712.2009.00646.x. PMID 20370749
- [Background] Shah A, Mosdossy G, McLeod S, Lehnhardt K, Peddle M, Rieder M. A blinded, randomized controlled trial to evaluate ketamine/propofol versus ketamine alone for procedural sedation in children. Ann Emerg Med. 2011 May;57(5):425-33.e2. doi: 10.1016/j.annemergmed.2010.08.032. Epub 2010 Oct 13. PMID 20947210
- [Background] Godambe SA, Elliot V, Matheny D, Pershad J. Comparison of propofol/fentanyl versus ketamine/midazolam for brief orthopedic procedural sedation in a pediatric emergency department. Pediatrics. 2003 Jul;112(1 Pt 1):116-23. doi: 10.1542/peds.112.1.116. PMID 12837876
- [Background] Kennedy RM, Porter FL, Miller JP, Jaffe DM. Comparison of fentanyl/midazolam with ketamine/midazolam for pediatric orthopedic emergencies. Pediatrics. 1998 Oct;102(4 Pt 1):956-63. doi: 10.1542/peds.102.4.956. PMID 9755272
- [Background] Messenger DW, Murray HE, Dungey PE, van Vlymen J, Sivilotti ML. Subdissociative-dose ketamine versus fentanyl for analgesia during propofol procedural sedation: a randomized clinical trial. Acad Emerg Med. 2008 Oct;15(10):877-86. doi: 10.1111/j.1553-2712.2008.00219.x. Epub 2008 Aug 27. PMID 18754820
- [Background] Chiaretti A, Ruggiero A, Barone G, Antonelli A, Lazzareschi I, Genovese O, Paiano S, Sammartino M, Maurizi P, Riccardi R. Propofol/alfentanil and propofol/ketamine procedural sedation in children with acute lymphoblastic leukaemia: safety, efficacy and their correlation with pain neuromediator expression. Eur J Cancer Care (Engl). 2010 Mar;19(2):212-20. doi: 10.1111/j.1365-2354.2008.01006.x. Epub 2009 May 21. PMID 19490010
- [Background] Tosun Z, Esmaoglu A, Coruh A. Propofol-ketamine vs propofol-fentanyl combinations for deep sedation and analgesia in pediatric patients undergoing burn dressing changes. Paediatr Anaesth. 2008 Jan;18(1):43-7. doi: 10.1111/j.1460-9592.2007.02380.x. PMID 18095965
- [Background] Bhatt M, Kennedy RM, Osmond MH, Krauss B, McAllister JD, Ansermino JM, Evered LM, Roback MG; Consensus Panel on Sedation Research of Pediatric Emergency Research Canada (PERC) and the Pediatric Emergency Care Applied Research Network (PECARN). Consensus-based recommendations for standardizing terminology and reporting adverse events for emergency department procedural sedation and analgesia in children. Ann Emerg Med. 2009 Apr;53(4):426-435.e4. doi: 10.1016/j.annemergmed.2008.09.030. Epub 2008 Nov 20. PMID 19026467